CLINICAL TRIAL: NCT01117974
Title: Neck Liposuction With Tumescent Anesthesia for the Treatment of Obstructive Sleep Apnea - A Pilot Study
Brief Title: Neck Liposuction for the Treatment of Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dennis West, Associate Professor of Dermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU17637
Record Dates: First submitted 2010-03-19; First posted 2010-05-06 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposuction (Experimental)
  Interventions: Procedure: liposuction of the neck

INTERVENTIONS:
Procedure: liposuction of the neck — Liposuction will be performed to the surgical endpoint (skin thickness in the suctioned areas similar to that of surrounding non-treated skin).

SUMMARY:
Liposuction, one of the most common cosmetic procedures performed in the United States, is a surgical technique used to reduce localized areas of excess subcutaneous fat. The neck is a common area of treatment, where liposuction reduces fat volume and neck size. We hypothesize that suctioned removal of fat of the neck will reduce the severity of obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years of age
* Subjects must have documented mild to moderate obstructive sleep apnea(OSA) syndrome within the last year from the Northwestern University Sleep Clinic
* Subjects must qualify as "very sleepy" on the Epworth Sleepiness Scale
* Females must have neck circumference of 16.0 cm or greater, and males must have neck circumference of 17.0 cm or greater
* Subjects must be a good candidates for neck liposuction as determined by the study physician
* Subjects must be in good health and is able to undergo the liposuction procedure

Exclusion Criteria:

* Pregnant or lactating female
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects dependent on blood thinners
* Subjects with bleeding diathesis
* Subjects with a history of poor wound healing, skin fragility, poor skin elasticity, or hypertrophic or keloidal scarring
* Subjects with a history of excessive surgeries on the neck in the area to be treated
* Subjects who are allergic to lidocaine or who have previously had an adverse reaction to epinephrine
* Subjects with non-apnea sleep disorders such as restless leg syndrome, insomnia, circadian rhythm disorders
* Subjects with chronic obstructive pulmonary disease
* Subjects with craniofacial abnormalities
* Subjects with hypoventilation
* Subjects with large tonsils/adenoids or an abnormal airway exam as determined by the study physician
* Subjects with an anatomical nasal obstruction
* Subjects who have a large tongue
* Subjects with severe cardiopulmonary risks as determined by the study physician
* Subjects who cannot complete an MRI
* Subjects who intend to pursue other treatments for OSA during the duration of this study
* Any previous and/or pending procedures at the treatment area or that may likely affect the treatment area
* Pending and/or anticipated major change in diet or exercise pattern in the six weeks following the last treatment
* Subjects with a Body Mass Index >35kg/m2
* Subjects treated with continuous positive airway pressure (CPAP) within one month of study enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | Baseline (0 weeks)
Change in the apnea-hypopnea index | 12 weeks

SECONDARY OUTCOMES:
Sleep-related quality of life | Baseline (Week 0)
Change in sleep-related quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yoo, MD, Principal Investigator — Northwestern University; Dennis P West, PhD, Principal Investigator — Northwestern University